CLINICAL TRIAL: NCT02013713
Title: French Observatory of Familial Hypercholesterolemia in Cardiology
Acronym: FH Care
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 12 449
Record Dates: First submitted 2013-12-06; First posted 2013-12-17 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Familial Hypercholesterolemia
Keywords: Cardiology; Family Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Family Hypercholesterolemia in cardiology

SUMMARY:
The Family Hypercholesterolemia remains poorly diagnosed disease with an outlet sometimes suboptimal care. However, the Family Hypercholesterolemia exposes patients concerned at increased cardiovascular risk.

The frequency of familial hypercholesterolemia in cardiologic is little studied and remains unknown, and there is little data on the profile of patients, diagnostic methods and management.

Main objectives:

* Establish a monitoring patients with hypercholesterolemia Family cardiology in France
* Characterize the Family hypercholesterolemia in cardiology, including assessing the frequency of the most severe forms, which are at higher cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* coronary patients
* who agreed to participate
* high LDL-c levels: * LDL-c> = 1.9g / l without lipid lowering treatment according to the diagnostic score of Family Hypercholesterolemia these coronary patients with LDL> 1.9g / l may possibly or probably be achieved Hypercholesterolemia Family.

or

* LDL-c> = 1.6g / l in lipid-lowering treatment, the reduction of LDL-c average expected under standard lipid-lowering therapy (statin alone) being 30-40% of these patients had therefore pretreatment levels greater than 2 g / l or greater than 2.5 g / l and may possibly or probably be achieved Family Hypercholesterolemia after the diagnostic score.

Exclusion Criteria:

* Expressed refusal to participate in the observatory
* Age ≤ 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is proposed to cardiology services hospitals. Aged 18 or more, seen in cardiology (USIC, Hospitalization, Consultation), who agreed to participate in the observatory, and coronary patients who have LDL-c levels
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Frequency of the Family Hypercholesterolemia in cardiology | 1 day
  Number of Family Hypercholesterolemia among patients with LDL-C> 1.9g / l without hypoglycemic treatment or> 1.6g / l in lipid-lowering therapy

CONTACTS AND LOCATIONS:
Locations (1):
- European Hospital Georges Pompidou, Paris, France

REFERENCES:
- [Background] Civeira F; International Panel on Management of Familial Hypercholesterolemia. Guidelines for the diagnosis and management of heterozygous familial hypercholesterolemia. Atherosclerosis. 2004 Mar;173(1):55-68. doi: 10.1016/j.atherosclerosis.2003.11.010. PMID 15177124